CLINICAL TRIAL: NCT02506140
Title: A Randomized, Open-label, Active-Controlled and Blinded-Endpoint Trial Comparing the Antiplatelet Effects of Ticagrelor Plus Aspirin Versus Clopidogrel Plus Aspirin in Chinese Patients With High-risk Transient Ischemic Attack or Minor Stroke.
Brief Title: Platelet Reactivity in Acute Non-disabling Cerebrovascular Events
Acronym: PRINCE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Beijing Municipal Science & Technology Commission (Other)
Responsible Party: Principal Investigator, Yongjun Wang, Executive Vice-President, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D151100002015001; 81322019 (Other Grant/Funding Number: National Natural Science Foundation of China)
Record Dates: First submitted 2015-07-19; First posted 2015-07-23 (Estimated); Last update posted 2020-07-24 (Actual); Status verified 2017-12

CONDITIONS: Stroke; Ischemic Attack, Transient
Keywords: minor stroke; transient ischemic attack; ticagrelor; clopidogrel; dual anti-platelet therapy; platelet reactivity
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient | interventions — Ticagrelor; Aspirin; Clopidogrel

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ticagrelor/ASA (Experimental): Drugs: Ticagrelor and Acetylsalicylic acid.
  Interventions: Drug: Ticagrelor and Acetylsalicylic acid
- Clopidogrel/ASA (Active Comparator): Drugs: Clopidogrel and Acetylsalicylic acid.
  Interventions: Drug: Clopidogrel and Acetylsalicylic acid

INTERVENTIONS:
Drug: Ticagrelor and Acetylsalicylic acid — This group will receive a 180 mg loading dose of ticagrelor on the day of randomization, followed by 90 mg twice/day ticagrelor from Day 2 to 3 months; combined with Aspirin given in a total dose of 100-300 mg on the first day, followed by 100 mg once/day from Day 2 to Day 21.
  Other Names: BRILINTA; Aspirin
  Arms: Ticagrelor/ASA
Drug: Clopidogrel and Acetylsalicylic acid — This group will receive a 300 mg loading dose of clopidogrel on the day of randomization, followed by 75 mg once/day clopidogrel from Day 2 to 3 months; combined with Aspirin given in a total dose of 100-300 mg on the first day, followed by 100 mg once/day from Day 2 to Day 21.
  Other Names: Plavix; Aspirin
  Arms: Clopidogrel/ASA

SUMMARY:
Ticagrelor is a reversible and direct-acting oral antagonist of the P2Y12 (Purinergic receptor P2Y, G-protein coupled, 12) receptor for adenosine diphosphate, which provides faster, greater, and more consistent P2Y12 inhibition than Clopidogrel in patients with acute coronary syndrome, irrespective of the genetic variants affecting Clopidogrel metabolism. It is still undefined whether combination therapy of Ticagrelor and Aspirin is more effective than Clopidogrel and aspirin for minor stroke and transient ischemic attack (TIA). The primary purpose of the PRINCE trial is to evaluate the anti-platelet effects of a 3-month regimen of ticagrelor initiated with 180 mg loading dose followed by 90 mg twice/day combined with aspirin 100 mg/day during first 21 days versus a 3-month regimen of clopidogrel initiated with 300 mg loading dose of followed by 75 mg/day combined with aspirin 100 mg/day during first 21 days when initiated within 24 hours of symptom onset in high-risk transient ischemic attack or minor stroke.

DETAILED DESCRIPTION:
The PRINCE trial is a prospective, randomized, multi-centre, open-label, active-controlled, blinded-endpoint trial (a PROBE design concerning clinical trial). A total of approximately 952 patients (40years≤Age<80years) with high-risk TIA (defined as an ABCD2 score ≥ 4 or the stenosis of offending vessel ≥ 50%) or minor ischemic stroke (defined as an NIHSS ≤ 3), who can be treated within 24 hours of symptom onset will be enrolled. Patients fulfilling all of the inclusion criteria and none of the exclusion criteria will be randomized 1:1 into two groups after offering informed content: 1) one group will receive a 180 mg loading dose of ticagrelor on the day of randomization, followed by 90 mg twice/day ticagrelor from Day 2 to 3 months; 2) the other group will receive a 300 mg loading dose of clopidogrel on the day of randomization, followed by 75 mg once/day clopidogrel from Day 2 to 3 months. Aspirin will be given in a total dose of 100-300 mg on the first day, followed by 100 mg once/day from Day 2 to Day 21 in the both groups. The primary objective is to assess the anti-platelet effects of Ticagrelor combined with Aspirin versus Clopidogrel combined with Aspirin in Chinese patients with high-risk TIA and minor stroke. The study consists of six visits including the day of randomization, 2 hours after the first anti-platelet agents, 24 hours after the first anti-platelet agents, Day 7+2days, Day 21±2days and Day 90±7days. Genomic DNA of all patients will be collected for genotyped. And the genetic variants affecting Clopidogrel metabolism will be analyzed. The antiplatelet effects will be analyzed in total subjects and genetic variants carriers. The trial is anticipated to complete in 18 months from the first subject recruitment , with 952 subjects recruited from 25 centres in China. A Data and Safety Monitoring Board (DSMB) will regularly monitor safety during the study. The trial has been approved by IRB(Institutional Review Board) /EC(Ethics Committee) in Beijing Tiantan hospital, Capital Medical University.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent.
2. Female or male aged≥ 40 years and <80 years.
3. Acute non-disabling ischemic stroke (NIHSS≤ 3 at the time of randomization) that can be treated with study drug within 24 hours of symptoms onset defined by the"last see normal"principle.
4. TIA (Neurological deficit attributed to focal brain ischemia, with resolution of the deficit within 24 hours of symptom onset), that can be treated with study drug within 24 hours of symptoms onset and with moderate-to-high risk of stroke recurrence (ABCD2 score ≥ 4 at the time of randomization or the stenosis of offending vessel ≥ 50%).

Exclusion Criteria:

1. Diagnosis of hemorrhage or other pathology, such as vascular malformation, tumor, abscess or other major non-ischemic brain disease (e.g., multiple sclerosis) on baseline head Computed Tomography (CT) or magnetic resonance imaging (MRI).
2. Isolated or pure sensory symptoms (e.g., numbness), isolated visual changes, or isolated dizziness/vertigo without evidence of acute infarction on baseline head CT or MRI.
3. Modified Rankin Scale Score > 2 at randomization (pre-morbid historical assessment)。
4. Contraindication to ticagrelor, clopidogrel or acetylsalicylic acid :

   * Known hypersensitivity
   * Severe renal or hepatic insufficiency
   * Severe cardiac failure, asthma
   * Hemostatic disorder or systemic bleeding
   * History of hemostatic disorder or systemic bleeding
   * History of drug-induced hematologic or hepatic abnormalities
   * Low white blood cell (<2 x10^9/L) or platelet count (<100 x10^9/L)
5. Clear indication for anticoagulation (presumed cardiac source of embolus, e.g., atrial fibrillation, ventricular aneurysm, prosthetic cardiac valves known, suspected endocarditis or other suspicion of cardioembolic pathology for TIA/stroke).
6. Continuous use of ticagrelor or clopidogrel over 5 days before randomization
7. Current treatment (last dose given within 10 days before randomization) with heparin therapy or anti coagulation therapy (e.g., warfarin; thrombin inhibitors such as dabigatran , argatroban, bivalirudin, ximelagatran; factor Xa inhibitors such as rivaroxaban, edoxaban, apixaban, betrixaban, tanexaban ; hirudin; unfractionated and low molecular weight heparins ).
8. Receipt of intravenous/ intra-arterial thrombolysis or mechanical thrombectomy within 24 hours prior to randomization.
9. History of intracranial hemorrhage or cerebral artery amyloidosis.
10. History of aneurysm (including intracranial aneurysm or peripheral aneurysms)
11. Diagnosis or of acute coronary syndrome.
12. History of asthma or COPD (chronic obstructive pulmonary disease).
13. High risk of bradyarrhythmia, such as sick sinus syndrome second-degree or third-degree atrioventricular block, bradycardia-related syncope without installed pacemaker.
14. History of uric acid nephropathy.
15. Anticipated requirement for long-term (>7 days) non-study anti-platelet drugs, or NSAIDs (nonsteroidal antiinflammatory drugs) affecting platelet function.
16. History of previous symptomatic non-traumatic intracerebral bleed at any time (asymptomatic microbleeds do not qualify), gastrointestinal (GI) bleed within the past 3 months, or major surgery within 30 days.
17. Qualifying TIA or minor stroke induced by angiography or surgery.
18. Planned or likely revascularization within the next 3 months.
19. Scheduled for surgery or interventional treatment requiring study drug cessation.
20. Severe non-cardiovascular comorbidity with life expectancy < 3 months.
21. Pregnancy or lactation, and women of childbearing age not practicing reliable contraception who do not have a documented negative pregnancy test.
22. Currently receiving an investigational drug or device.
23. Participation in another clinical study with an investigational product during the last 30 days.
24. Inability of the patient to understand and/or comply with study procedures and/or follow-up, in the opinion of the Investigator.
25. Hematocrit (Hct) < 30%

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 675 (Actual)
Dates: Start 2015-08; Primary Completion 2017-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
High on-treatment platelet reactivity (HOPR) defined as P2Y12 reaction unit (PRU)> 208 measured by VerifyNow® assay at 90 days | 90 days

SECONDARY OUTCOMES:
HOPR at 90 days in subjects carrying genetic variants which affected Clopidogrel metabolism. | 90 days
  HOPR defined as P2Y12 reaction unit (PRU)> 208 measured by VerifyNow® assay
New vascular events defined as any event of the following: Any stroke (ischemic or hemorrhage). | 90 days, 6 months, 1 year
  All the new vascular events will be assessed by at least two neurologists based on neuroimaging and clinical feature. When there was disagreement, a third senior neurologist was consulted to reach a consensus decision.
New composite clinical vascular events (ischemic stroke/ hemorrhagic stroke/TIA/ myocardial infarction/ vascular death) as a cluster. | 90 days, 6 months, 1 year
  All the new composite clinical vascular events will be assessed by at least two neurologists based on laboratory examination, imaging and clinical feature. When there was disagreement, a third senior neurologist was consulted to reach a consensus decision.
High on-treatment platelet reactivity defined as PRU> 208 measured by VerifyNow® assay. | 2hours, 24 hours, 7 days
High on-treatment platelet reactivity defined as Aspirin reactivity unit (ARU)> 555 measured by VerifyNow® assay. | 7 days
HOPR defined as Maximum Amplitude-adenosine diphosphate (MA-ADP)>47 measured by Thrombelastography Platelet Mapping Assay (TEG) using the inducer of adenosine diphosphate. | 90 days
Residual platelet reactivity defined as the value of PRU. | 2hours, 24 hours, 7 days, 90 days
Residual platelet reactivity defined as the value of Aspirin reaction unit (ARU). | 7days
Residual platelet reactivity defined as the value of MA-ADP. | 7days, 90 days
Residual platelet reactivity defined as the value of Maximum Amplitude- acetylsalicylic acid (MA-AA) measured by TEG. | 7days
Residual platelet reactivity change from baseline in PRU. | 2hours, 24 hours, 7 days, 90 days
Residual platelet reactivity change from baseline in ARU. | 7 days
The inhibition of platelet aggregation (IPA) measured by VerifyNow® assay. | 2hours, 24 hours, 7 days, 90 days
The TEG-platelet inhibition(TPI)measured by TEG. | 7 days, 90 days
Platelet inhibition change from baseline in IPA. | 2hours, 24 hours, 7 days, 90 days
Platelet inhibition change from baseline in TPI. | 7 days, 90 days
Residual platelet reactivity detected by AspirinWorks. | 7days
Residual platelet reactivity detected by PL Platelet Analyser (SINNOWA®). | 7days, 90days
Modified Rankin Scale score changes (continuous) and dichotomized at percentage with score 0-2 vs. 3-6. | 90 days, 6 months, 1 year
Further efficacy exploratory analysis:Impairment (changes in NIHSS scores at 90 days, 6 months, 1 year follow-up) | 90 days, 6 months, 1 year
Further efficacy exploratory analysis:Quality of Life (The EuroQol-5D 3 level version[EQ-5D-3L]scale). | 90 days, 6 months, 1 year
Major bleed (PLATO definition), including fatal/life-threatening and other. | 90 days, 6 months, 1 year
  The PLATO(Platelet Inhibition and Patient Outcomes) definition of fatal/life-threatening of major bleed is any one of the following: Fatal, Intracranial, Intrapericardial bleed with cardiac tamponade, Hypovolaemic shock or severe hypotension due to bleeding and requiring pressors or surgery, Clinically overt or apparent bleeding associated with a decrease in hemoglobin(Hb) of more than50 g/L, Transfusion of 4 or more units (whole blood or packed red blood cells [PRBCs]) for bleeding. The PLATO definition of other of major bleed is any one of the following:Significantly disabling (eg. intraocular with permanent vision loss), Clinically overt or apparent bleeding associated with a decrease in Hb of 30 g/L to 50 g/L, Transfusion of 2-3 units (whole blood or PRBCs) for bleeding.
Intracranial hemorrhagic events. | 90 days, 6 months, 1 year
  Intracranial hemorrhagic events is assessed by brain computed tomography (CT) or gradient recalled echo (GRE) T2 star weighted MRI.
Total mortality. | 90 days, 6 months, 1 year
  All deaths reported post-randomization will be recorded and adjudicated. Deaths will be subclassified by the adjudication committee as cardiovascular or non-cardiovascular.

CONTACTS AND LOCATIONS:
Locations (25):
- China (25):
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - The Second People's Hospital of Shenzhen, Shenzhen, Guangdong
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - North China University of Science And Technology Affiliated Hospital, Tangshan, Hebei
  - Tangshan Gongren Hospital, Tangshan, Hebei
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Wuhan Brain Hospital,General Hospital of The Yangtze River Shipping, Wuhan, Hubei
  - Union Hospital,Tongji Medical College,Huazhong University of Science and Technology, Wuhan, Hubei
  - Wuhan No.1 Hospital, Wuhan, Hubei
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Northern Jiangsu People's Hospital,Clinical Medical School,YangZhou University, Yangzhou, Jiangsu
  - General Hospital of Shenyang Military, Shengyang, Liaoning
  - The Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - General Hospital of TISCO, Taiyuan, Shanxi
  - Taizhou First People's Hospital,Huangyan Hospital of Wenzhou Medical University, Taizhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Wenzhou Hospital of integrated Chinese and Western medicine, Wenzhou, Zhejiang
  - Aviation General Hospital of China Medical University, Beijing
  - Beijing Tian Tan Hospital, Capital Medical University, Beijing
  - Dongfang Hospital Beijing University of Chinese Medicine, Beijing
  - The First Hospital of Fangshan District,Beijing, Beijing
  - Daping Hospital,Third Military Medical University, Chongqing
  - Renji Hospital,Shanghai Jiao Tong University School of Medicine, Shanghai
  - Tianjin Huanhu Hospital, Tianjin

REFERENCES:
- [Derived] Yang Y, Chen W, Pan Y, Yan H, Meng X, Liu L, Wang Y, Wang Y. Ticagrelor Is Superior to Clopidogrel in Inhibiting Platelet Reactivity in Patients With Minor Stroke or TIA. Front Neurol. 2020 Jun 10;11:534. doi: 10.3389/fneur.2020.00534. eCollection 2020. PMID 32587571
- [Derived] Yang Y, Chen W, Meng X, Liu L, Wang Y, Pan Y, Wang Y. Impact of smoking on platelet function of ticagrelor versus clopidogrel in minor stroke or transient ischaemic attack. Eur J Neurol. 2020 May;27(5):833-840. doi: 10.1111/ene.14171. Epub 2020 Mar 8. PMID 32052517
- [Derived] Wang Y, Chen W, Lin Y, Meng X, Chen G, Wang Z, Wu J, Wang D, Li J, Cao Y, Xu Y, Zhang G, Li X, Pan Y, Li H, Zhao X, Liu L, Lin J, Dong K, Jing J, Johnston SC, Wang D, Wang Y; PRINCE Protocol Steering Group. Ticagrelor plus aspirin versus clopidogrel plus aspirin for platelet reactivity in patients with minor stroke or transient ischaemic attack: open label, blinded endpoint, randomised controlled phase II trial. BMJ. 2019 Jun 6;365:l2211. doi: 10.1136/bmj.l2211. PMID 31171523
- [Derived] Wang Y, Lin Y, Meng X, Chen W, Chen G, Wang Z, Wu J, Wang D, Li J, Cao Y, Xu Y, Zhang G, Li X, Pan Y, Li H, Liu L, Zhao X, Wang Y; PRINCE Protocol Steering Group. Effect of ticagrelor with clopidogrel on high on-treatment platelet reactivity in acute stroke or transient ischemic attack (PRINCE) trial: Rationale and design. Int J Stroke. 2017 Apr;12(3):321-325. doi: 10.1177/1747493017694390. Epub 2017 Jan 1. PMID 28381198